CLINICAL TRIAL: NCT02755753
Title: A Multicenter, Randomized, Double-blinded, Placebo-controlled Pilot Study to Evaluate the Efficacy and Safety of Rebamipide as an Adjuvant Regimen to Heal erosIve Reflux Esophagitis (REPAIR)
Brief Title: A Study to Evaluate REbamiPide as an Adjuvant Regimen to Heal erosIve Reflux Esophagitis
Acronym: REPAIR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: YongChan Lee (Other)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor-Investigator, YongChan Lee, Professor, Severance Hospital
Organization: Severance Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 037-OTC-1201i
Record Dates: First submitted 2015-09-02; First posted 2016-04-29 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Gastroesophageal Reflux
Keywords: Rebamipide
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Lansoprazole; rebamipide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Study Group (Experimental): 1. Lanston® (lansoprazole) 30 mg, 1 capsule, PO, qd, 30 min before breakfast
  2. Mucosta® (rebamipide) 100 mg, 1 tablet, PO, tid, 30 minutes before breakfast, lunch and dinner
  Interventions: Drug: Lansoprazole; Drug: Rebamipide
- Control Group (Placebo Comparator): 1. Lanston® (lansoprazole) 30 mg, 1 capsule, PO, qd, 30 min before breakfast
  2. Mucosta®-placebo (rebamipide-placebo), 1 tablet, PO, tid, 30 minutes before breakfast, lunch and dinner
  Interventions: Drug: Lansoprazole; Drug: Rebamipide-placebo

INTERVENTIONS:
Drug: Lansoprazole — Oral administration of Lanston® (lansoprazole) 30 mg, 1 capsule, PO, qd, 30 min before breakfast
  Other Names: Lanston
Drug: Rebamipide — Oral administration of Mucosta (rebamipide) 100 mg, 1 tablet, PO, tid, 30 minutes before breakfast, lunch, and dinner
  Other Names: Mucosta
  Arms: Study Group
Drug: Rebamipide-placebo — Oral administration of Mucosta®-placebo, 1 tablet, PO, tid, 30 minutes before breakfast, lunch and dinner
  Other Names: Mucosta-placebo
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate whether Rebamipide facilitate the healing of inflamed mucosa as an adjuvant regimen in erosive reflux esophagitis (ERE).

DETAILED DESCRIPTION:
1. To evaluate whether Rebamipide facilitate the healing of inflamed mucosa as an adjuvant regimen in erosive reflux esophagitis patients
2. To evaluate the safety of rebamipide as an adjuvant regimen in erosive reflux esophagitis (ERE)

ELIGIBILITY:
Inclusion Criteria:

1. Male/female patients aged 20 to 70 at the time of writing an informed consent.
2. Subjects who were diagnosed with Erosive Reflux Esophagitis (ERE) using Los Angeles (LA) classification grade A~D, confirmed by endoscopy.
3. The subjects regardless of presence of ERE symptom (i.e., symptomatic ERE or asymptomatic ERE).

   For symptomatic ERE, the subject must have one or more symptoms of the followings: acid regurgitation, heartburn, epigastric pain, cough, hoarseness, globus pharyngis, atypical chest pain.
4. Subjects who have consented to participate in this clinical study by signing an informed consent form.

Exclusion Criteria:

1. Patients with known hypersensitivity to any component of Lanston® and/or Mucosta® formulations.
2. Other concurrent organic upper gastroesophageal disease in endoscopy (i.e., drug-induced esophagitis, viral esophagitis, Mallory-Weiss syndrome, peptic ulcer disease, malignancies) and patients who was diagnosed with Barrett's esophagus.
3. History of abdominal surgery that can affect gastrointestinal motility (except appendectomy and hysterectomy).
4. History of upper gastrointestinal bleeding or obstruction.
5. Patients administrated with any drugs that can affect the efficacy of study regimen (proton pump inhibitors, revaprazan, prokinetics, H2-blockers, etc.) within 2 weeks (however, 4 weeks for PPIs) prior to enrollment and/or those who are required of NSAIDs, anti-coagulants, anti-cholinergics, prostaglandin E, corticosteroids, and anti-depressants treatment during the study period.
6. History of pancreatobiliary disease (except asymptomatic gallbladder stone), inflammatory bowel disease, cirrhotic liver disease, chronic kidney disease.
7. Pregnant, nursing, and childbearing potential women who is unwilling to effective contraception; for example, oral contraceptives, hormonal methods, placement of an intrauterine device (IUD) or intrauterine system (IUS), barrier methods (i.e., condom or occlusive cap with spermicidal foam/gel/film/cream/suppository), male sterilization, and true abstinence.
8. History of psychological disorder, alcoholics, and drug abuser.
9. Blood test results of hemoglobin (Hb) ≤ 10.0 g/dL, platelets ≤ 50,000 /µL, total WBCs ≤ 4,000/µL or ≥ 10,000/µL, and with serum test results showing the levels of AST, ALT, ALP, BUN, and creatinine exceeding twice the normal range of respective institution.
10. Patients who previously underwent another clinical survey within 4 weeks.
11. History of major medical disease that can affect general condition and other patients deemed not eligible for this study by investigators.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Endoscopic healing rate | 4 weeks
  The ratio of the endoscopically completely healed (normal or minimal change) patients per groups

SECONDARY OUTCOMES:
Histologic change | 4 weeks
  Histologic change defined with Hematoxylin and eosin (H&E) stain
Change in inflammatory cytokines | 4 weeks
  Change in the tissue level of Platelet activating factor (PAF) and Interleukin-8 (IL-8)
Time to complete symptom relief | every 2 week, up to 4 week
  Interval between inital medication and the first time of symptom relief judged by subject's diary
Overall symptom relief | every 2 week, up to 4 week
  The proportion of relieved subjects at the end of treatment
Adverse events profile | every 2 week, up to 4week
  patient's symptoms, physical findings, abnormal laboratory values, vital signs, and ECG findings

CONTACTS AND LOCATIONS:
Overall Officials: Yong Chan Lee, MD, PhD, Principal Investigator — Severance Hospital, Yonsei University Health System; Seong Woo Jeon, MD, PhD, Principal Investigator — Kyungpook National University Medical Center; Su Jin Hong, MD, PhD, Principal Investigator — Soonchunhyang University Buchen Hospital; Kyung Ho Song, MD, Master, Principal Investigator — Konyang University Hospital; Shiming Yang, MD, PhD, Principal Investigator — Xinqiao Hospital of Chongqing
Locations (5):
- Yang Shiming, Chongqing, Chongqing Municipality, China
- South Korea (4):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Kyungpook National University Medical Center, Daegu
  - Konyang University Hospital, Daejeon
  - Severance Hospital, Yonsei University Health System, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chai J, Jamal MM. Esophageal malignancy: a growing concern. World J Gastroenterol. 2012 Dec 7;18(45):6521-6. doi: 10.3748/wjg.v18.i45.6521. PMID 23236223
- [Background] Vakil N, van Zanten SV, Kahrilas P, Dent J, Jones R; Global Consensus Group. The Montreal definition and classification of gastroesophageal reflux disease: a global evidence-based consensus. Am J Gastroenterol. 2006 Aug;101(8):1900-20; quiz 1943. doi: 10.1111/j.1572-0241.2006.00630.x. PMID 16928254
- [Background] Peery AF, Dellon ES, Lund J, Crockett SD, McGowan CE, Bulsiewicz WJ, Gangarosa LM, Thiny MT, Stizenberg K, Morgan DR, Ringel Y, Kim HP, DiBonaventura MD, Carroll CF, Allen JK, Cook SF, Sandler RS, Kappelman MD, Shaheen NJ. Burden of gastrointestinal disease in the United States: 2012 update. Gastroenterology. 2012 Nov;143(5):1179-1187.e3. doi: 10.1053/j.gastro.2012.08.002. Epub 2012 Aug 8. PMID 22885331
- [Background] Wong RK, Yeoh KG, Gwee KA, Tay HW, Ho KY. Validation of structured scoring using the LA classification for esophagitis and endoscopically suspected Barrett's esophagus in a tertiary Asian endoscopy center. J Gastroenterol Hepatol. 2009 Jan;24(1):103-6. doi: 10.1111/j.1440-1746.2008.05680.x. Epub 2008 Dec 1. PMID 19054260
- [Background] Dent J, El-Serag HB, Wallander MA, Johansson S. Epidemiology of gastro-oesophageal reflux disease: a systematic review. Gut. 2005 May;54(5):710-7. doi: 10.1136/gut.2004.051821. PMID 15831922
- [Background] Kang JY. Systematic review: geographical and ethnic differences in gastro-oesophageal reflux disease. Aliment Pharmacol Ther. 2004 Oct 1;20(7):705-17. doi: 10.1111/j.1365-2036.2004.02165.x. PMID 15379831
- [Background] Kim KM, Cho YK, Bae SJ, Kim DS, Shim KN, Kim JH, Jung SW, Kim N. Prevalence of gastroesophageal reflux disease in Korea and associated health-care utilization: a national population-based study. J Gastroenterol Hepatol. 2012 Apr;27(4):741-5. doi: 10.1111/j.1440-1746.2011.06921.x. PMID 21916988
- [Background] Song JH, Chung SJ, Lee JH, Kim YH, Chang DK, Son HJ, Kim JJ, Rhee JC, Rhee PL. Relationship between gastroesophageal reflux symptoms and dietary factors in Korea. J Neurogastroenterol Motil. 2011 Jan;17(1):54-60. doi: 10.5056/jnm.2011.17.1.54. Epub 2011 Jan 26. PMID 21369492
- [Background] Lee SJ, Song CW, Jeen YT, Chun HJ, Lee HS, Um SH, Lee SW, Choi JH, Kim CD, Ryu HS, Hyun JH. Prevalence of endoscopic reflux esophagitis among Koreans. J Gastroenterol Hepatol. 2001 Apr;16(4):373-6. doi: 10.1046/j.1440-1746.2001.02464.x. PMID 11354273
- [Background] Hwang JK, Kim J, Hong SG, Jung SJ, Joo MK, Lee BJ, Park JJ, Kim JS, Bak YT. [A prospective multicenter study on the prevalence and symptoms of erosive reflux esophagitis in secondary and tertiary hospitals in Korea]. Korean J Gastroenterol. 2009 May;53(5):283-91. doi: 10.4166/kjg.2009.53.5.283. Korean. PMID 19458464
- [Background] Kim BJ, Cheon WS, Oh HC, Kim JW, Park JD, Kim JG. Prevalence and risk factor of erosive esophagitis observed in Korean National Cancer Screening Program. J Korean Med Sci. 2011 May;26(5):642-6. doi: 10.3346/jkms.2011.26.5.642. Epub 2011 Apr 21. PMID 21532855
- [Background] Li YM, Du J, Zhang H, Yu CH. Epidemiological investigation in outpatients with symptomatic gastroesophageal reflux from the Department of Medicine in Zhejiang Province, east China. J Gastroenterol Hepatol. 2008 Feb;23(2):283-9. doi: 10.1111/j.1440-1746.2007.05045.x. Epub 2007 Jul 20. PMID 17645475
- [Background] Shaw MJ, Crawley JA. Improving health-related quality of life in gastro-oesophageal reflux disease. Drugs. 2003;63(21):2307-16. doi: 10.2165/00003495-200363210-00003. PMID 14524732
- [Background] Kovacs TO, Freston JW, Haber MM, Atkinson S, Hunt B, Peura DA. Long-term quality of life improvement in subjects with healed erosive esophagitis: treatment with lansoprazole. Dig Dis Sci. 2010 May;55(5):1325-36. doi: 10.1007/s10620-009-0871-8. Epub 2009 Jul 7. PMID 19582579
- [Background] Howden CW, Chey WD. Gastroesophageal reflux disease. J Fam Pract. 2003 Mar;52(3):240-7. PMID 12620183
- [Background] Lee JH, Cho YK, Jeon SW, Kim JH, Kim NY, Lee JS, Bak YT; Korean Society of Neurogastroenterology and Motility. [Guidelines for the treatment of gastroesophageal reflux disease]. Korean J Gastroenterol. 2011 Feb;57(2):57-66. doi: 10.4166/kjg.2011.57.2.57. Korean. PMID 21350318
- [Background] Kovacs TO, Freston JW, Haber MM, Hunt B, Atkinson S, Peura DA. Long-term efficacy of lansoprazole in preventing relapse of erosive reflux esophagitis. Dig Dis Sci. 2009 Aug;54(8):1693-701. doi: 10.1007/s10620-009-0769-5. Epub 2009 Mar 7. PMID 19267194
- [Background] Yoshida N, Kamada K, Tomatsuri N, Suzuki T, Takagi T, Ichikawa H, Yoshikawa T. Management of recurrence of symptoms of gastroesophageal reflux disease: synergistic effect of rebamipide with 15 mg lansoprazole. Dig Dis Sci. 2010 Dec;55(12):3393-8. doi: 10.1007/s10620-010-1166-9. Epub 2010 Mar 3. PMID 20198424
- [Background] Hatlebakk JG, Berstad A. Lansoprazole 15 and 30 mg daily in maintaining healing and symptom relief in patients with reflux oesophagitis. Aliment Pharmacol Ther. 1997 Apr;11(2):365-72. doi: 10.1046/j.1365-2036.1997.144320000.x. PMID 9146777
- [Background] Lancaster GA, Dodd S, Williamson PR. Design and analysis of pilot studies: recommendations for good practice. J Eval Clin Pract. 2004 May;10(2):307-12. doi: 10.1111/j..2002.384.doc.x. PMID 15189396
- [Background] Hongo M. Minimal changes in reflux esophagitis: red ones and white ones. J Gastroenterol. 2006 Feb;41(2):95-9. doi: 10.1007/s00535-006-1775-4. PMID 16568367
- [Background] Kusano M, Ino K, Yamada T, Kawamura O, Toki M, Ohwada T, Kikuchi K, Shirota T, Kimura M, Miyazaki M, Nakamura K, Igarashi S, Tomizawa M, Tamura T, Sekiguchi T, Mori M. Interobserver and intraobserver variation in endoscopic assessment of GERD using the "Los Angeles" classification. Gastrointest Endosc. 1999 Jun;49(6):700-4. doi: 10.1016/s0016-5107(99)70285-3. PMID 10343212
- [Background] Fiocca R, Mastracci L, Milione M, Parente P, Savarino V; Gruppo Italiano Patologi Apparato Digerente (GIPAD); Societa Italiana di Anatomia Patologica e Citopatologia Diagnostica/International Academy of Pathology, Italian division (SIAPEC/IAP). Microscopic esophagitis and Barrett's esophagus: the histology report. Dig Liver Dis. 2011 Mar;43 Suppl 4:S319-30. doi: 10.1016/S1590-8658(11)60588-4. PMID 21459338
- [Result] Holzheimer RG, Mannick JA, editors. Surgical Treatment: Evidence-Based and Problem-Oriented. Munich: Zuckschwerdt; 2001. Available from http://www.ncbi.nlm.nih.gov/books/NBK6880/ PMID 21028753